CLINICAL TRIAL: NCT00954213
Title: A One-year Prospective Follow-up Study of a DIR/ Floortime Parent Training Intervention for Pre-school Children With Autistic Spectrum Disorders
Brief Title: A Study of a Developmental,Individual-Difference,Relationship-Bases/Floortime Intervention for Children With Autistic
Acronym: DIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Associate Professor Dr. Kingkaew Pajareya,M.D., Rehabilitation Medicine, Siriraj Hospital, Bangkok, Thailand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206/2551(EC1)
Record Dates: First submitted 2009-08-04; First posted 2009-08-07 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DIR/Floortime parent intervention (Experimental)
  Interventions: Behavioral: DIR/Floortime parent intervention

INTERVENTIONS:
Behavioral: DIR/Floortime parent intervention — Parent will be trained to observe their autistic child's cues, follow their child's lead and techniques to enhance his/her development.

SUMMARY:
Thirty eight autistic spectrum disorder children age 2-6 years recruited into the study. The new treatment intervention is based on the DIR Model. Parents will be coached at the start and then every 3-4 months for 1 year. Outcome will be measured at the first session and at the end of the study using Functional Emotional Assessment Scale and Childhood Autism Rating Scales, Functional Emotional Level, and parent satisfaction rating.

Hypothesis of the study: Children who get additional treatment of DIR/floortime show much improvement in climbing the developmental "ladder" and declining in the autistic behaviors.

ELIGIBILITY:
Inclusion Criteria:

* clinical criteria for Autistic Disorders according to DSM IV
* child is 2 - 6 years of age

Exclusion Criteria:

* children with additional medical diagnosis (e.g., genetic syndromes, diagnosed hearing impairment, diagnosed visual impairment or seizures)
* children who are geographically inaccessible for follow-up visits
* their parents are not literate or known chronic psychiatric or physical illness in the parents

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The Functional Emotional Assessment Scale (FEAS) Ratings (the child part) | 1 year

SECONDARY OUTCOMES:
The Childhood Autism Rating Scale (CARS) Clinical rating of the children (6 point scale related to Greenspan's six Functional Development Level -FDL) Satisfaction of the effectiveness of the intervention of their child (Six-point Likert scale) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kingkaew Pajareya, MD, Principal Investigator — Rehabilitation Medicine, Siriraj Hospital, Bangkok, Thailand
Locations (1):
- Kingkaew Pajareya, Bangkoknoi, Bangkok, Thailand